CLINICAL TRIAL: NCT04702139
Title: Use of the "Game-Ready" Splint for Better Recovery in Primary Total Shoulder Arthroplasty
Acronym: game-ready
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A02470-39
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2023-09

CONDITIONS: Shoulder Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with game-ready splint (Active Comparator): Installation of the Game-Ready splint immediately after surgery for 12 hours. They will then be put on the standard splint which they will keep for 2 weeks as for the other group but without ice packs.
  Interventions: Device: shoulder arthroplastis
- patient with standard splint (Placebo Comparator): Placement of a standard splint immediately after surgery for 2 weeks with ice packs to be used for an average of 8 days.
  Interventions: Device: shoulder arthroplastis

INTERVENTIONS:
Device: shoulder arthroplastis — - Group (Treatment): Placement of the Game-Ready splint immediately after surgery for 12 hours. They will then be put on the standard splint which they will keep for 2 weeks as for the other group but without ice packs.
  Arms: patient with game-ready splint
Device: shoulder arthroplastis — - Group (Control): Placement of a standard splint immediately after surgery for 2 weeks with ice packs to be used for an average of 8 days.
  Arms: patient with standard splint

SUMMARY:
The aim of the study is to compare the level of postoperative pain after fitting the Game Ready splint, at 48 hours versus that observed with fitting a standard splint

ELIGIBILITY:
Inclusion Criteria:

1. First-line reverse prosthesis
2. Without prosthetic history
3. Patient who has given his consent to participate in the observational study after being informed by the surgeon
4. Patient living in France and able to answer the questionnaire alone.
5. Subject affiliated to a social security scheme or beneficiary of such a scheme
6. Lack of participation in another clinical study

Exclusion Criteria:

1. Minor patient
2. Major subject protected by law, under curatorship or tutorship
3. Anterior prosthesis
4. Infection
5. Parkinson's, degenerative neurological disease
6. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
the level of postoperative pain following the installation of the Game Ready | 9 months
  Visual Analog Score for pain

SECONDARY OUTCOMES:
risk of stiffness | up to 9 months
  Physicians Global Assessment to measure risk of stiffness
occurrence of hematoma, edema | up to 9 months
  Physicians Global Assessment to measure the occurrence of hematoma, edema
length of hospitalization | up to 24 hours
  Physicians Global Assessment to measure the length of hospitalisation
evolution of mobility | up to 9 months
  Simple shoulder test, subjective shoulder value, and American Shoulder and Elbow Surgeons Shoulder Score
the time limit for returning to a possible professional activity | up to 3 months
  Physicians Global Assessment to measure quality of life

CONTACTS AND LOCATIONS:
Overall Officials: philippe VALENTI, DOCTOR, Principal Investigator — Clinique Bizet
Locations (1):
- Bizet Clinic, Paris, France

IPD SHARING:
Plan to Share IPD: No